CLINICAL TRIAL: NCT02789384
Title: Prognostic Value of the CINSARC (Complexity Index in Sarcoma) Signature and Correlation With Chemotherapy Efficacy in Soft-tissue Sarcomas. A Biomarker Study. (NEOSarcomics )
Brief Title: CINSARC Signature and Correlation With Hemotherapy Efficacy in Soft-tissue Sarcomas. A Biomarker Study.
Acronym: NEOSarcomics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IB 2015-07
Record Dates: First submitted 2016-04-29; First posted 2016-06-03 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Soft-tissue Sarcomas
Keywords: soft-tissue sarcomas; CINSARC; biomarker; efficacy; pronostic
MeSH Terms: conditions — Sarcoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Procedure/Surgery (Experimental): Newly obtained biopsy if applicable and blood samples collection according to the usual medical practices.
  Interventions: Other: Procedure/Surgery

INTERVENTIONS:
Other: Procedure/Surgery — Procedure/Surgery: Newly obtained biopsy if applicable and Blood samples collection.
  For each patient:
  * Frozen and paraffin embedded tumor material (archival or new biopsy) will be obtained for genetic profiling
  * Blood samples will be obtained for genetic profiling and assessment of markers.
  The classification as CINSARC will be performed for each patient. Patients should be treated by neoadjuvant anthracycline-based chemotherapy. Chemotherapy regimen must contain at least doxorubicin (dose range: 60 -75 mg/m²) and ifosfamide (dose range: 2.5-3g/m²) to be delivered on a 21-days cycle basis up to 6 cycles prior surgery. After neoadjuvant chemotherapy completion, patients will be treated by surgery followed or not by radiotherapy.
  All patients should be managed according to the usual medical practices.

SUMMARY:
This is a prospective observational biomarker study including patients with non-metastatic, soft-tissue sarcomas (STS) for whom neoadjuvant chemotherapy is considered as the best option by the multidisciplinary sarcoma team of one of the participating centers.

DETAILED DESCRIPTION:
Even when retrospective statistical identification for a biomarker has been achieved, the ultimate proof of its usefulness in the clinic still requires prospective evidence. Our prospective study aims to validate the prognosis value of the CINSARC signature in a prospective way. Moreover, the neoadjuvant setting is an ideal one to identify molecular predictive factors of sensitivity to chemotherapy by correlating tumor response with genetic profile of STS. Moreover, molecular profiling of treatment-refractory tumor cells may reveal alterations that are associated with drug resistance, metastatic recurrence and disease progression. The identifications of such factors in the neoadjuvant setting may help to improve the management of STS patients in the adjuvant and metastatic settings

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed soft-tissue sarcoma by central review, except if the diagnosis was already confirmed by the RRePS (Réseau de Référence en Pathologie des Sarcomes et des Viscères) Network,
2. Available archived frozen tumor tissue sample or patient consenting to undergo a biopsy of the tumour for research purpose,
3. Non-metastatic disease, for which the use of chemotherapy to "downstage" the sarcoma prior to surgery, is assumed to result in better local tumor control by the multidisciplinary sarcoma team of one of the French reference centers involved in this study,
4. Age ≥ 18 years,
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1,
6. Measurable disease according to RECIST v1.1 outside any previously irradiated field,
7. Neoadjuvant anthracycline-based chemotherapy proposed as the best option by the multidisciplinary sarcoma team of one of the French reference centers involved in this study,
8. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
9. Voluntarily signed and dated written informed consents prior to any study specific procedure,
10. Patients with a social security in compliance with the French Law relating to biomedical research (Article 1121-11 of French Public Health Code).

Exclusion Criteria:

1. Pathological diagnosis different from a soft-tissue sarcoma,
2. Histological subtypes: well-differentiated liposarcoma, alveolar soft-part sarcoma, dermatofibrosarcoma protuberans, clear-cell sarcoma, rhabdomyosarcoma,
3. Previous treatment for the sarcoma,
4. Contra-indication precluding the administration of chemotherapy as assessed by the investigator,
5. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
6. Previous enrolment in the present study,
7. Pregnant or breast feeding women,
8. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of antitumor activity of neoadjuvant anthracycline based chemotherapy. Efficacy will be defined based on complete response, partial response and stable disease observed during treatment following RECIST v1.1 criteria. | participants will be followed for the duration of treatment, an expected average of 6-months

SECONDARY OUTCOMES:
Efficacy of neoadjuvant anthracycline based chemotherapy in terms of proportion of tumour cells identified on the surgical specimen | an expected average of 6 months
Association of the CINSARC signature and histological response based on the proportion of tumour cells identified on the surgical specimen | an expected average of 6 months
Patient's classification by CINSARC signature. Patients will be classified as either low risk CINSARC or high risk | 6 months
Metastasis-free survial is defined following recent guidelines for the definition of survival endpoints in sarcoma trials (Bellera et al. Annals Oncol 2014. | 3 years
3 -year Overall Survial (OS) defined as the time from study treatment initiation to death (of any cause). | 3 years
Histological response is defined using both 3 histological parameters: proportion of recognizable tumor cells, fibrosis and necrosis in the surgical specimen. | an expected average of 6 months
Identification of molecular mechanisms involved in intrinsic resistance to chemotherapy by correlating the transcriptome data with response to chemotherapy. | an expected average of 6 months
Adverse events related to the biopsy procedure will be graded using the common toxicity criteria from the NCI v4.0. | during 7 days after biopsy

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - AP-HM _ Hôpital de la Timone, Marseille
  - Institut de Cancérologie de l'Ouest, Nantes
  - Institut Curie, Paris
  - Institut Claudius Regaud - IUCT-0, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guegan JP, El Ghazzi N, Vibert J, Rey C, Vanhersecke L, Coindre JM, Toulmonde M, Spalato Ceruso M, Peyraud F, Bessede A, Italiano A. Predictive value of tumor microenvironment on pathologic response to neoadjuvant chemotherapy in patients with undifferentiated pleomorphic sarcomas. J Hematol Oncol. 2024 Oct 23;17(1):100. doi: 10.1186/s13045-024-01614-w. PMID 39444039